CLINICAL TRIAL: NCT06551974
Title: Development of a Guided Self-help Mobile App to Improve Treatment Outcome for Individuals Suffering From Eating Disorders
Brief Title: INTERconNEcT-Eds: a Guided Self-help Mobile App to Improve Outcome in Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: University of Catanzaro (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Gianluca Lo Coco, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prot. P202237PFB
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Eating Disorder Symptom; Eating Disorders; Eating Behavior
Keywords: eating disorders; guided self-help; online intervention; peer mentoring; tailored interventions; interpersonal group; therapeutic alliance
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior | interventions — adenylate isopentenyltransferase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Guided self-help plus IPT (Experimental): The participants will have access to self-help materials (workbook and videoclips), forum groups (interactional materials), online interpersonal group sessions for 8 weeks. Participants will use self-help materials through a mobile app and online platform. Regarding anorexic symptoms and behaviours, the self-help material will focus on the topics of the New Maudsley model. Further modules will cover the ED overeating problems and the interpersonal difficulties related to EDs.
  The weekly online forum group is focused on interactional material that will be delivered weekly through a synchronous 1-hour mobile chat with a peer mentor (a recovered influencer). Each session lasts 60 minutes and is themed following the structure of the video-clips materials.
  Finally, 90-minute interpersonal group sessions will be led online by clinicians with an expertise in the treatment of eating disorders.
  Interventions: Behavioral: Guided self-help plus IPT
- Treatment-as-usual (Active Comparator): Treatment as usual will vary between centres and this will impact the effect size of the intervention (Ayling et al., 2015). We will therefore conduct structured interviews with clinicians at each study site to clarify the nature of treatment as usual at each centre. We will also use an adapted form of the Client Service Receipt Inventory (a well-established tool used in health economics) to track the amount of treatment received over the year (Beecham & Knapp, 1992). The inventory will be administered at 8-week and 3-month, to measure patients' service usage.
  Interventions: Behavioral: TAU
- Guided self-help (Experimental): The participants will have access to self-help materials (workbook and videoclips), and forum groups (interactional materials). Participants will use self-help materials through a mobile app and online platform. Regarding anorexic symptoms and behaviours, the self-help material will focus on the topics of the New Maudsley model. Further modules will cover the ED overeating problems and the interpersonal difficulties related to EDs.
  The weekly online forum group is focused on interactional material that will be delivered weekly through a synchronous 1-hour mobile chat with a peer mentor (a recovered influencer). Each session lasts 60 minutes and is themed following the structure of the video-clips materials.
  Interventions: Behavioral: Guided self-help
- No treatment (No Intervention): The no-treatment control condition includes participants with sub-threshold eating symptoms who attend regular visits with their own primary care physician. In this context, it is important that participants, interested to take part to the study, offered number or contact of the own primary care physician in case of an illness worsening.

INTERVENTIONS:
Behavioral: Guided self-help plus IPT — The participants allocated in the intervention GSH arm will have access to self-help materials (workbook and videoclips), forum groups (interactional materials), online interpersonal group sessions for 8 weeks. The proposed online GSH will be adapted from two online interventions developed and tested with people with eating disorders by the Eating Disorders Research Unit team at King's College London, with a cooperation of the University of Palermo research team (Cardi et al., 2020). The GSH will include self-help materials, i.e. a written workbook and a library of 74 brief video-clips with the goal of providing psychoeducation about eating disorders and interpersonal difficulties and describing and modelling the use of helpful strategies to reverse abnormal eating behaviours. Participants will also attend a weekly online forum with interactional materials, and an online interpersonal group session.
  Arms: Guided self-help plus IPT
Behavioral: Guided self-help — The participants allocated in the intervention GSH arm will have access to self-help materials (workbook and videoclips), forum groups (interactional materials), online interpersonal group sessions for 8 weeks. The proposed online GSH will be adapted from two online interventions developed and tested with people with eating disorders by the Eating Disorders Research Unit team at King's College London, with a cooperation of the University of Palermo research team (Cardi et al., 2020). The GSH will include self-help materials, i.e. a written workbook and a library of 74 brief video-clips with the goal of providing psychoeducation about eating disorders and interpersonal difficulties and describing and modelling the use of helpful strategies to reverse abnormal eating behaviours.
  Arms: Guided self-help
Behavioral: TAU — The Treatment as Usual is the usual or routine care provided to participants in the outpatient setting.
  Arms: Treatment-as-usual

SUMMARY:
Eating disorders (EDs) are psychiatric illnesses characterised by pathological eating behaviours, ranging from protracted undereating to recurrent loss of control over eating. Based on the transdiagnostic approach, EDs are triggered and maintained by interpersonal distress and difficulties to manage negative emotions. Thus, interpersonal skills have been implicated as important targets for change in the treatment. In this project, we will adopt digital technologies to improve treatment adherence and outcome of individuals with EDs, by testing the effectiveness of an online self-help program delivered through a mobile app. Specifically, this project aims to establish if an online personalized self-help approach is feasible and effective in ameliorating eating disorder symptoms and distress. We planned to conduct two randomised controlled trials to test the effectiveness of online guided self-help (GSH) in two different settings: (1) the community, and (2) the outpatient setting. This is to establish at which stage of treatment this approach is most helpful. Across studies, we will recruit 242 individuals aged ≥18 years with ED symptoms and/or a proper diagnosis of EDs (DSM-5). During eight weeks period, GSH will be available to participants both on a website and a new-developed smartphone app and consists of written materials and brief video-clips, a weekly chat based forum group and an online interpersonal group session. Guidance in forum groups will be facilitated by non-specialist help-care providers (i.e., peer mentors); whereas experienced mental health providers will lead the online group sessions. Participant's interpersonal distress will be assessed at intake to personalize guidance in the group, by addressing dysfunctional interpersonal characteristics which can be associated with ED symptoms. Participants will also complete a weekly working alliance measure to examine whether the quality of relationship with mentor predicts clients' level of clinical change.

Regarding the outpatient setting, the first aim is to assess if GSH intervention is effective to improve the following primary outcome for patients with ED diagnosis: 1) overall psychological distress. In the community setting, the study aims to examine if GSH is effective to improve the following primary outcomes for individuals with self-reported ED symptoms: 1) overall psychological distress; 2) first contact with clinical services to manage their dysfunctional eating behaviors.

DETAILED DESCRIPTION:
Despite the disabling nature of eating disorders, many individuals with EDs do not receive appropriate mental health care. Recently, the use of eHealth technology has been proposed as a potentially effective alternative to traditional, inperson treatment delivery for those with EDs. Specifically, self-help programs include the use of materials, such as books, workbooks and videoclips, to empower patients through information and skills to cope with the illness. Guided self-help adds the element of guidance to the use of these materials.

The project aims to exploit the use of highly scalable and inclusive digital technologies (i.e., mobile app and online GSH) to improve the transdiagnostic understanding of EDs and their psychological treatment. Online GSH will be developed based on pre-existing UK-based model of intervention (RecoveryMANTRA and ECHOMANTRA) and will be adapted to Italian young adults through the introduction of a smartphone app aimed to monitor and support individuals to treatment. This project aims to establish at what stage of illness the evidence-based interventions used are most valued and beneficial to individuals. Therefore, online GSH will be tested in two different settings and clinical context: (1) the outpatient setting for those reporting a diagnosis of ED; and (2) the community setting for people reporting symptoms of eating disorders who are not receiving psychological treatment. GSH translated for delivery through smartphone app may be one solution towards reducing treatment gap for people with ED who do not still receive a proper support, fostering awareness and motivation to start treatment as well as an augmenting strategy to improve clinical outcomes for patients undergoing routine treatment delivered by clinical services.

Primary aims: Regarding the outpatient setting, the first aim is to assess if GSH intervention is effective to improve the following primary outcome for patients with ED diagnosis: 1) overall psychological distress. Secondary outcomes are: 1) eating disorder psychopathology; 2) interpersonal distress; 3) quality of life; 4) motivation for treatment; 5) emotion dysregulation; 6) Body Mass Index, 7) satisfaction with treatment, at the end of the 8-week intervention and 3-month follow-up compared to the control condition.

In the community setting, the study aims to examine if GSH is effective to improve the following primary outcome for individuals with symptoms of disordered eating: 1) overall psychological distress; Secondary outcomes are: 1) eating disorder psychopathology; 2) interpersonal distress; 3) quality of life; 4) motivation for treatment; 5) emotion dysregulation, 6) Body Mass Index, 7) satisfaction with treatment, 8) first contact with clinical services to manage their dysfunctional eating behaviors, at the end of the 8-week GSH and at 3-month follow-up compared to the control condition. Secondary aims: A secondary aim is to determine the extent to which the working alliance with clinicians delivering weekly online group guidance is associated with clients' clinical changes on a session-by-session basis during the intervention. Given the difficult nature of building a strong therapeutic alliance with ED patients (Warren, Crowley, Olivardia & Schoen, 2008), an increased willingness to trust in clinician during the online GSH may be a basis for increased treatment involvement and symptomatic improvement.

Study 1. The first study is a multicentric RCT where participants with a proper diagnosis of eating disorders will be recruited at the Eating Disorders Unit of the University Hospital of Catanzaro and Padova. The aim of this RCT is to answer to the question: "Does online guided self-help through mobile app for eating disorders provided in addition to TAU improve overall psychological distress, eating disorder psychopathology, BMI, interpersonal distress, quality of life, motivation for treatment, emotion dysregulation, satisfaction with treatment compared to treatment as usual alone (outpatient treatment) among young people with a diagnosis of eating disorders?".

Participants will be randomized to one of two groups: (1) online guided self-help + treatment as usual (EDs standard treatment by participating centres) or (2) treatment as usual only). After completing informed consent and baseline questionnaires, participants will be randomised to the intervention or control group, using a web-based randomisation tool. Randomization will take place in blocks, in size of 16 participants, with a 1:1 allocation ratio to ensure a random allocation of 8 participants in each group per time. The participants allocated in the intervention arm will get access to self-help materials (workbook and videoclips), forum groups (interactional materials) and online interpersonal group sessions for 8 weeks.

Study 2. In this RCT, participants will be recruited from the community through advertisements posted in the psychoeducation Instagram profile "Dicci Come Aiutarti" (Albano et al. 2023). The aim of this RCT is to answer to the question: "Does online guided self-help through mobile app for eating disorders improve overall psychological distress as well as eating disorder psychopathology, BMI, interpersonal distress, quality of life, motivation for treatment, emotion dysregulation, satisfaction with treatment and service use, compared to a no treatment condition?". A secondary aim of this trial is to evaluate if during the ongoing trial or at the end of the intervention (8 weeks) participants start a clinical intervention in a specialized service to manage their eating difficulties.

Participants will be randomized to one of two groups: (1) online guided self-help (without online interpersonal sessions) or (2) TAU (only GP consultation). After completing informed consent and baseline questionnaires, participants will be randomised to the intervention or control group using a web-based randomisation tool, with a 1:1 allocation ratio.

Guided self-help intervention. The proposed 8-week online GSH will be adapted from two online interventions developed and tested with people with eating disorders by the Eating Disorders Research Unit team at King's College London, with a cooperation of the University of Palermo research team (Cardi et al., 2020). The GSH will include self-help materials, i.e. a written workbook and a library of 74 brief video-clips with the goal of providing psychoeducation about eating disorders and interpersonal difficulties and describing and modelling the use of helpful strategies to reverse abnormal eating behaviours. Participants will use self-help materials through a mobile app and online platform, which will be developed and implemented by the Tech Digit Easy s.r.l., a company leader in the design and development of E-health services and devices which has been cooperating with the Research Unit of the University of Palermo for 2 years. Regarding anorexic symptoms and behaviours, the self-help material will focus on the topics of the New Maudsley model. Therefore, participants will get the chance to work on six main areas related to EDs maintenance factors. On the other hand, further modules will cover the ED overeating behaviors through the Italian translation of the manual Getting Better Bite by Bite: A Survival Kit for Sufferers of Bulimia Nervosa and Binge Eating Disorders (Schmidt, Treasure & Alexander, 2012). Finally, a module on interpersonal difficulties related to EDs will be provided to all participants as a transdiagnostic maintenance illness factor to be addressed (Rieger, Van Buren, Bishop, Tanofsky-Kraff, Welch, & Wilfley, 2010; Wilfley et al., 2002).

A further service offered through the mobile app will be the chance to get access to a weekly online forum group (interactional material) aimed to foster the adherence to the self-help program and the use of online materials. A focus on motivation to change, instilling hope on the recovery, will be promoted through motivational interviewing framework and the lived experience of influencers who recovered from an EDs (collaborators of #DCA). This additional interactional material will be delivered weekly through a synchronous 1-hour mobile chat with a peer mentor (a recovered influencer from an EDs) and a low experienced professional (graduated students in psychology). Each session lasts 60 minutes and is themed following the structure of the patient video-clips materials.

In this project, interpersonal group sessions (IPT) involve 90-minute weekly online sessions (Murphy et al., 2012). Group sessions will be led by clinicians with a good expertise in the treatment of eating disorders. The interpersonal group sessions could be attended by those participants enrolled in the study and recruited from clinical centres with a proper diagnosis of eating disorder. The interpersonal group sessions will be delivered through a zoom link available in the online platform. A group of 6-8 participants, diagnosed with various eating disorders including AN, BN, and BED, will be included with the aim of addressing the interpersonal difficulties related to nutrition and eating management.

Statistical Analysis Power analysis: An a-priori sample size was estimated using G*Power, based on previous research findings (e.g., Cardi et al., 2020 Traviss-Turner et al., 2017). Considering a mixed design factorial ANOVA, a statistical power of (1 - β) = .90, alpha level of .05, a small effect size (Cohen's f = .10) in mean improvement for outcome variables, and medium to high stability of the outcomes across time points (r= .60), the power analysis suggested a sample to include 86 subjects per group, with a total of 172 participants in the study 1. An a-priori sample size was estimated using G*Power, based on previous research findings (e.g., Linardon, Shatte, Rosato & Fuller-Tyszkiewicz, 2022). Considering a mixed design factorial ANOVA, a statistical power of (1 - β) = .80, a two-tailed alpha level and a small effect size (Cohen's f = .10) in mean improvement for outcome variables, and medium to high stability of the outcomes across time points (r = .60), the power analysis suggested a sample to include 35 subjects per group, with a total of 70 participants in the study 2.

For first aim: Univariate analyses of variance will be used to compare the intervention and control arms on the clinical outcomes. All analyses will be based on the intention-to-treat approach. Missing data will be imputed using multiple imputation based upon the Markov chain Monte Carlo method and maximum likelihood imputation based upon the Expectation-Maximization (EM) algorithm. Results will be compared across the two methods. Linear Mixed-effects Models applying an intent-to-treat approach will be used to compare the intervention arm to the control group in terms of both primary and secondary outcomes. Effect sizes will be calculated using Cohen's d.

For the secondary aim: The random intercepts cross-lagged panel model will assess the bidirectional association between working alliance and post-session weekly outcomes (EDE-Q, CORE-10 etc). The random intercept in the model removes between-person variance (i.e., Level 2) such that the lagged relationships in the cross-lagged model characterize within-person change over time. Three fit indices will be used to evaluate the fit of the model: the comparative fit index (CFI), root mean square error of approximation (RMSEA), and standardized root mean square residual (SRMR). Two models will be estimated, one with the auto-correlation and the cross-lagged paths freely estimated, and a second model with the auto-correlation and the cross-lagged paths constrained to be equal across time periods.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for study 1 are: (1) >18 years, (2) with a clinician-formulated diagnosis of eating disorder (i.e., anorexia nervosa, bulimia nervosa, binge eating disorder) or Other Specified Feeding or Eating Disorder based on the criteria of the DSM-5-TR, (3) having started TAU within 12 months; (4) with access to Internet connection through a mobile device, (5) Italian speaking.

The inclusion criteria for study 2 are: (1) >18 years, (2) a score > 2.77 on the Eating Disorders Examination Questionnaire, (3) attending no treatment for eating disorder symptoms but reporting a regular monitoring by their own primary care physician (GP), 4) with access to Internet connection through a mobile device, (4) Italian speaking.

Exclusion Criteria:

For both study 1and 2: acute psychosis, clinical depression or suicidal ideation, pregnancy, use of medication that might influence eating behavior, neurological and visual impairment and Intellectual disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM): | Baseline, end-of-treatment (8 weeks), and 3-month follow-up.
  The CORE-OM is a 34-item validate, self-report scale (of which 25% are reverse items) assessing global distress of the subject across 4 domains: [Well-being (4 items); Functioning (12 items); Problems/symptoms (12 items); Risk (to self and to others) (6 items)] over the last week.
  Items are answered on the same five-point scale (0-4) ranging from 'not at all' to 'most or all the time'. Overall, the measure is problem scored (i.e. higher scores indicate more problems). Scores are reported as means across items that give a 'pro-rated' score if there are incomplete responses.

SECONDARY OUTCOMES:
Change from baseline in the Eating Disorder Examination Questionnaire | Baseline, 8 weeks, and 3-month follow-up.
  Questionnaire (EDE-Q 6.0): it is a self-report scale assessing eating disorder psychopathology and behaviors. The questionnaire is made up of 22 items, rated on a 7-point from 0 to 6. Higher scores reflecting greater severity or frequency. It also provides frequency data on key behavioral features of eating disorders, in terms of the number of episodes of the behavior over the preceding 28 days, and the number of days on which the behavior has occurred. Items are grouped into 4 subscales: restraint, weight concern, shape concern and eating concern.
Change from baseline in the Inventory of Interpersonal Problems | Baseline, 8 weeks, and 3-month follow-up.
  The IIP-32 is a self-report scale 32-item inventory of distressing interpersonal behaviours the respondent identifies as "hard to do" (i.e., behavioural inhibitions) or "does too much" (i.e., behavioural excesses) on a 0 (not at all) to 4 (extremely) Likert scale. It provides an overall score and 8 subscale scores: (Domineering/Controlling, Vindictive/Self-centered, Cold/distant, Socially inhibited, Nonassertive, Overly accommodating, Self-sacrificing, Intrusive needy).
  Higher scores in each scale indicate the presence of interpersonal difficulties.
Change from baseline in the Autonomous and Controlled Motivation for Treatment Questionnaire | Baseline, 8 weeks, and 3-month follow-up.
  The ACMTQ consists of two subscales assessing autonomous and controlled motivation for treatment through 12-items on a seven-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate a stronger endorsement of the motivation type.
Change from baseline in the Difficulties in Emotion Regulation Scale | Baseline, 8 weeks, and 3-month follow-up.
  The Difficulties in Emotion Regulation Scale (DERS) is a 5-point self-report instrument measuring emotion regulation problems. The 36 items (of which 11 are reverse items) asks respondents how they relate to their emotions in order to produce scores on the following subscales: non acceptance of emotional responses, difficulty engaging in goal-directed behaviour, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, lack of emotional clarity. Higher scores suggest greater problems with emotion regulation.
Change from baseline in the Client Satisfaction Questionnaire | Baseline, 8 weeks, and 3-month follow-up.
  The Client Satisfaction Questionnaire is an eight-item self-report measure aimed at measuring participant satisfaction with treatment, with a Likert scale ranging from 0 to 6. Higher scores indicate better outcome. In the present study, the researchers adapted the CSQ to include one additional question to measure satisfaction with online-based treatment.

OTHER OUTCOMES:
Change from baseline in the EQ-5D-5L | Baseline, 8 weeks, and 3-month follow-up.
  The EQ-5D-5L descriptive system includes ﬁve dimensions: mobility (MO), self-care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD). Each dimension is articulated into ﬁve severity levels: no problems, slight problems, moderate problems, severe problems, extreme problems. The EQ-5D questionnaire also includes a visual analogue scale (EQ VAS) on which participants indicated their self-rated health at the time between 0 (worst imaginable health) and 100 (best imaginable health).
Change from baseline in Body Mass Index | Baseline, weekly, 8 weeks, and 3-month follow-up.
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
  BMI categories:
  Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9 Obesity = BMI of 30 or greater
Change from baseline in use of care services | Baseline, 8 weeks, and 3-month follow-up.
  Participant's Service Use (PSU). Participants in study 2 will indicate the type of care service used in the last 6 weeks and the number of days they have used a service in the last 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Lo Coco, Principal Investigator — University of Palermo; Cristina Segura-Garcia, Study Director — University of Catanzaro
Locations (1):
- Outpatient Unit for Clinical research and Treatment of Eating Disorders. University Hospital Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of the main outcome article, after deidentification (text, tables and figures).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Lo Coco G, Albano G, Gullo S, Cardi V, Segura-Garcia C. The feasibility, acceptability and clinical impact of a guided self-help mobile intervention (INTERconNEcT-EDs) for individuals with eating disorders: protocol for two multicenter randomized controlled trials. J Eat Disord. 2025 Jun 23;13(1):119. doi: 10.1186/s40337-025-01320-z. PMID 40551261